CLINICAL TRIAL: NCT06465264
Title: Efficacy and Safety of Allisartan Isoproxil/Amlodipine in Patients With Essential Hypertension Uncontrolled With Amlodipine or Allisartan Isoproxil: A Phase III, Multicenter, Randomized, Double-blind, Parallel-controlled, 52-week Clinical Study
Brief Title: To Assess Allisartan Isoproxil/Amlodipine in Patients With Essential Hypertension Uncontrolled With Amlodipine or Allisartan Isoproxil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL0107A103
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Essential Hypertension
Keywords: Allisartan Isoproxil; Amlodipine; Essential hypertension; Systolic BP; Diastolic BP
MeSH Terms: conditions — Essential Hypertension | interventions — allisartan isoproxil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind treatment (Week 4~Week 16):
  Open-label period(Week 16~ Week 56):
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Allisartan Isoproxil/Amlodipine group 1 (Experimental): Patients will be treated with one Allisartan Isoproxil/Amlodipine (240 mg/5 mg) tablet and one placebo of Amlodipine during the double-blind period (Week 4~Week 16) and one Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Interventions: Drug: Allisartan Isoproxil/Amlodipine group 1
- Amlodipine group 1 (Active Comparator): Patients will be treated with one Amlodipine (5 mg) tablet and one placebo of Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the double-blind period (Week 4~Week 16) and one Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Interventions: Drug: Amlodipine group 1
- Allisartan Isoproxil/Amlodipine group 2 (Experimental): Patients will be treated with one Allisartan Isoproxil/Amlodipine (240 mg/5 mg) tablet and one placebo of Allisartan Isoproxil tablet during the double-blind period (Week 4~Week 16) and one Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Interventions: Drug: Allisartan Isoproxil/Amlodipine group 2
- Allisartan Isoproxil group 2 (Active Comparator): Patients will be treated with one Allisartan Isoproxil (240 mg) and one placebo of Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the double-blind period (Week 4~Week 16) and one Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Interventions: Drug: Allisartan Isoproxil group 2

INTERVENTIONS:
Drug: Allisartan Isoproxil/Amlodipine group 1 — One Allisartan Isoproxil/Amlodipine (240 mg/5 mg) tablet and one placebo of Amlodipine during the double-blind period (Week 4~Week 16).
  One Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Arms: Allisartan Isoproxil/Amlodipine group 1
Drug: Amlodipine group 1 — One Amlodipine (5 mg) tablet and one placebo of Allisartan Isoproxil/Amlodipine during the double-blind period (Week 4~Week 16).
  One Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Arms: Amlodipine group 1
Drug: Allisartan Isoproxil/Amlodipine group 2 — One Allisartan Isoproxil/Amlodipine (240 mg/5 mg) tablet and one placebo of Allisartan Isoproxil (240 mg) during the double-blind period (Week 4~Week 16).
  One Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Arms: Allisartan Isoproxil/Amlodipine group 2
Drug: Allisartan Isoproxil group 2 — One Allisartan Isoproxil (240 mg) and one placebo of Allisartan Isoproxil/Amlodipine (240 mg/5 mg) during the double-blind period (Week 4~Week 16).
  One Allisartan Isoproxil/Amlodipine(240 mg/5 mg) tablet during the open-label period(Week 16~ Week 56) once daily.
  Arms: Allisartan Isoproxil group 2

SUMMARY:
The main objective of the study will be to assess the efficacy and safety of Allisartan Isoproxil/Amlodipine (240 mg/5 mg) in patients with mild to moderate essential hypertension uncontrolled after 4-week treatment with Amlodipine besylate（5 mg) or Allisartan Isoproxil (240 mg).

DETAILED DESCRIPTION:
Amlodipine belongs to the calcium channel blocker (CCB) class of drugs, which acts as an antihypertensive agent mainly via blocking calcium channels on the vascular smooth muscle cells to dilate blood vessels.

Allisartan Isoproxil belongs to the ARB class of drugs, which can effectively exert antihypertensive effects.

The combination of dihydropyridine CCBs and ARBs exerts synergistic antihypertensive effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old with mild to moderate essential hypertension;
* Untreated patients (either newly diagnosed essential hypertension or those patients with a history of hypertension but have not been taking any antihypertensive drugs for at least 2 weeks before the first visit) must have an office msSBP ≥ 150 mmHg and < 180 mmHg and DBP<110 mmHg;
* Patients who had not received regular treatment with Amlodipine Besylate (5 mg/day) (less than 4 weeks of medication intake or a history of missing doses for 5 or more days within the 4 weeks before screening) with the mean sitting blood pressure of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg;
* Patients currently receiving other antihypertensive agents (non-study medications for at least 2 weeks prior to screening) with the mean sitting blood pressure of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg, and the clinician determined that it was appropriate to switch to Amlodipine Besylate (5 mg/day);
* Patients who have been stably treated with Amlodipine Besylate (5 mg/day) for at least 4 weeks with the mean sitting blood pressure of 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg. During randomization for the double-blind treatment period, mean sitting blood pressure should be 140 mmHg≤ SBP <180 mmHg and DBP<110 mmHg;
* Participants enrolled in the ambulatory blood pressure monitoring (ABPM) study should have 24-hour mean ambulatory blood pressure ≥130/80 mmHg after 4 weeks of monotherapy treatment;

Exclusion Criteria:

* Patients with secondary hypertension;
* Patients with msSBP ≥180 mmHg and/or msDBP≥110 mmHg, or with hypertensive emergency or hypertensive urgency.
* Patients with history of heart failure (New York Heart Association (NYHA) Functional Classification class III and IV), acute coronary syndrome, percutaneous coronary intervention, or other serious heart diseases (such as cardiogenic shock, moderate or severe heart valvular disorders, atrioventricular block second or third degree, bradycardia (with a heart rate <50 beats per minute), severe arrhythmias) in the past 6 months.
* Patients with history of severe cerebrovascular diseases (such as hypertensive encephalopathy, cerebrovascular injury, stroke, transient ischemic attack) in the past 6 months.
* Patients with aortic aneurysm, aortic dissection, or dissecting aneurysm.
* Patients with renal artery stenosis or severe renal insufficiency (Cr>1.5 times the upper limit of normal).
* Patients with blood potassium >5.5 mmol/L.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 499 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure after 12 weeks of randomized, double-blind treatment | Baseline, week 12
  Twenty-four hour mean msSBP will be performed at baseline and week 12 of double-blind treatment

SECONDARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 12 weeks of randomized, double-blind treatment | Baseline, week 12
  Twenty-four hour mean msDBP will be performed at baseline and week 12 of double-blind treatment
Change from baseline in mean sitting systolic blood pressure and mean sitting diastolic blood pressure after 4 and 8 weeks of randomized, double-blind treatment | Baseline, week 4, week 8
  Twenty-four hour mean msSBP will be performed at baseline and week 4, week 8 of double-blind treatment
The proportion of responders to antihypertensive treatment after 12 weeks of randomized, double-blind treatment | Week 12
  Responders is the ratio of the number of participants achieving SBP/DBP<140/90 mmHg or a reduction from baseline of >20 mmHg in mean systolic blood pressure and or >10 mmHg in mean diastolic blood pressure to the total number of participants in each group
The proportion of patients meeting the mean sitting blood pressure target after 4, 8, and 12 weeks of randomized, double-blind treatment | Week 4, week 8, week 12
  Sitting blood pressure target is SBP/DBP<140/90 mmHg

OTHER OUTCOMES:
The proportion of patients meeting the mean sitting blood pressure target after 20 weeks of extended treatment | Week 36
  Sitting blood pressure target is SBP/DBP<140/90 mmHg
The proportion of patients meeting the mean sitting blood pressure target at the end of treatment | Week 56
  Sitting blood pressure target is SBP/DBP<140/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Xinchun Yang, Ph.D, Principal Investigator — Beijing Chaoyang Hospital, Capital Medical University City:Beijing
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chi H, Zhang X, Ma S, Pan G, Lian X, Chen Y, Pei H, Liu Z, Lin X. Efficacy and Safety of Allisartan Isoproxil/Amlodipine in Patients With Essential Hypertension Uncontrolled by Amlodipine: A Phase III, Multicenter, Double-Blind, Parallel-Group, Randomized Controlled Trial. J Clin Hypertens (Greenwich). 2025 Jan;27(1):e14955. doi: 10.1111/jch.14955. PMID 39821945